CLINICAL TRIAL: NCT05308433
Title: Cybersickness imAgiNg Olfactory Evocation
Acronym: CANOE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Cécile RUMEAU, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A02854-37
Record Dates: First submitted 2022-03-04; First posted 2022-04-04 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Healthy
Keywords: fMRI
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Device: Functional MRI; Other: Virtual Reality: control; Other: Virtual Reality: experimental

INTERVENTIONS:
Device: Functional MRI — The volunteer will have to imagine the smells evoked by different visual aids. This task will be carried out during 2 acquisition runs of about 10 minutes each. The volunteer should note (on a scale from 1 to 4) the pleasantness of the smell evoked.
  Other Names: fMRI
Other: Virtual Reality: control — The volunteer will be immersed in a virtual maritime environment with nauseating characteristics. In the center of the maritime scene, it will be visible the black outlines of a frame. Every minute, the volunteer will be asked to verbalize the level of his general condition via the Fast Motion Sickness Scale (1 to 20).
  Other Names: VR control
Other: Virtual Reality: experimental — The volunteer will be immersed in a virtual maritime environment with nauseating characteristics. The visual support inserted in the center of the virtual scene will be the one defined as being the most facilitator of the olfactory imagination during the fMRI examination. The volunteer will be asked to concentrate on the smell evoked by this support. Every minute, the volunteer will be asked to verbalize the level of his general condition via the Fast Motion Sickness Scale (1 to 20).
  Other Names: VR experimental

SUMMARY:
The aim of this study is to, using fMRI, compare brain activations during olfactory imagery induced by different visual supports (words, pictures, colors and colored arrangements) in healthy subjects.

This will allow us to choose the best olfactory imagery facilitator and to assess its effect on cybersickness.

ELIGIBILITY:
Inclusion Criteria:

* to be of French nationality who has always lived in metropolitan France;
* to be right-handed person;
* to be enrolled in a social security plan;
* to be able to understand the instructions given;
* to have underwent a pre-inclusion medical examination;
* to give a written consent;
* Person with a strong capacity for olfactory imagination: having obtained a score strictly below 2.5 on the fVOIQ olfactory imagination questionnaire.

Exclusion Criteria:

* to have an inability to read French;
* to be recognized as a synesthete;
* to have a professional activity requires intense olfactory activity;
* to have a partial or total loss of smell (hyposmia, anosmia);
* to have qualitative smell disorders (carcosomia, hyperosmia, phantosmia, parosmia);
* to have smell disorders of neurological, post-traumatic or neurodegenerative origin;
* to have uncorrected or poorly corrected visual disturbances;
* to have vestibular disorder diagnosed;
* any contraindication to MR examination (active medical device, ferromagnetic foreign body, pregnancy, morbid obesity, claustrophobia, … );
* subject under a measure of legal protection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Comparison of cerebral activations between the different supports mediating the olfactory imagination during the execution of the fMRI tasks. | Baseline (J0)
  The cerebral activations between the different supports mediating the olfactory imagination will be compared in terms of localization and intensity of the variations of the BOLD signal during the execution of the fMRI tasks.

SECONDARY OUTCOMES:
Determination of the visual support allowing the strongest olfactory imagination during the fMRI by subjective evaluations using two 4-level Likert scales. | Baseline (J0)
  Subjective evaluations will be carried out using two 4-level Likert scales.
Determination of the visual support allowing the strongest olfactory imagination during the fMRI test by the cerebral activations in areas recognized for their implications in the olfactory imagination. | Baseline (J0)
  The cerebral activations will be measured by the intensity of the variations of the BOLD signal during the execution of the fMRI tasks.
Description of the evolution of the cardiac activity during olfactory imagination tasks in fMRI. | Baseline (J0)
  The cardiac activity will be evaluated by the R-wave interval. The cardiac activity will be recorded via the ECG during olfactory imagination tasks in fMRI.
Description of the evolution of the respiratory activity during olfactory imagination tasks in fMRI. | Baseline (J0)
  The respiratory activity will be evaluated by the respiratory rate. The respiratory activity will be recorded via the respiratory belt during olfactory imagination tasks in fMRI.
Evaluation of the state of discomfort in virtual reality by measuring the cardiac activity. | Baseline (J0) and 6 months maximum after J0 (V1)
  Cardiac activity will be evaluated by the R-wave interval. Cardiac activity during immersion will be recorded by the cardio-respiratory belt.
Evaluation of the state of discomfort in virtual reality by the "Simulator Sickness Questionnaire" (SSQ) before and after immersion. | Baseline (J0) and 6 months maximum after J0 (V1)
  The participant will answer to the "Simulator Sickness Questionnaire" (SSQ) before and after immersion (minimum=0 and maximum=235,62). A higher score means a more severe discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France

REFERENCES:
- [Background] Fantin L, Ceyte H, Ramdane-Cherif Z, Jacquot M, Hossu G. French Vividness of Olfactory Imagery Questionnaire: A Potential Tool for Diagnosing Olfactory Loss by Assessing Olfactory Imagery? Front Psychol. 2020 Dec 21;11:606667. doi: 10.3389/fpsyg.2020.606667. eCollection 2020. PMID 33408672